CLINICAL TRIAL: NCT04541654
Title: Li-Fraumeni & TP53: Understanding and Progress (LiFT UP)
Brief Title: Li-Fraumeni & TP53 (LiFT UP): Understanding and Progress
Acronym: LiFT_UP
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); City of Hope Medical Center (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Judy E. Garber, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 20-226; R01CA242218 (NIH)
Record Dates: First submitted 2020-08-25; First posted 2020-09-09 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Li-Fraumeni Syndrome; TP53 Gene Mutation; Hereditary Cancer Syndrome; Clonal Hematopoiesis; Mosaicism
Keywords: Li-Fraumeni Syndrome; TP53 Gene Mutation (Variant); Hereditary Cancer Syndrome; Clonal Hematopoiesis; Mosaicism
MeSH Terms: conditions — Li-Fraumeni Syndrome; Neoplastic Syndromes, Hereditary | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Salivary DNA, Hair Follicle Specimens, Tumor or normal Tissue Specimens, Other Specimens*
  *Donation by participants of deceased family member's pathology specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Variant in the TP53 Gene in blood or saliva: Variant in the TP53 gene found on a blood or saliva test, have a relative with a variant in the TP53 gene, or because participant meets genetic testing criteria for Li-Fraumeni Syndrome (LFS) based on personal or family cancer history
  Interventions: Genetic: Data and Specimen Collection

INTERVENTIONS:
Genetic: Data and Specimen Collection — * Provide research team and access to relevant medical records
  * Answer short questionnaires periodically
  * Consider consenting to other optional parts of the research such as:
  * Providing up to 3 tubes (15ml) of blood at or near the time of consent, as approved by treating physician (optional).
  * Provide a saliva sample (optional).
  * Provide eyebrow hairs for analysis of DNA from the bulb (15-20 eyebrow plucks) (optional).
  * Provide permission for obtainment of stored tissue specimens from cancer or pre-cancer surgeries or biopsies from the pathology departments where they have been stored (optional).
  * Consider inviting relatives to join the study (optional).

SUMMARY:
The purpose of this research study is to learn more about variants in the TP53 gene both associated with Li-Fraumeni Syndrome (LFS), a hereditary cancer risk condition, and TP53 variants found in the blood for other reasons (e.g. ACE/CHIP and mosaicism).

DETAILED DESCRIPTION:
This research study looks to enroll as many people with LFS or TP53 gene variants as possible in order to:

* Better estimate cancer risks in individuals with TP53 variants or LFS, which is a rare condition.
* Learn the range of cancer risks linked to TP53 variants to help individuals and families to improve our ability to counsel patients and families about cancer risks more accurately.
* Improve opportunities for cancer prevention, early detection, and treatment.
* Learn more about the meaning of TP53 variants in the blood that are not inherited (e.g. ACE/CHIP and mosaicism).

Study procedures will include:

* Collecting information from the participant's medical record and short questionnaires.
* Collecting blood, saliva, eyebrow hair and tumor tissue samples (optional).
* Sharing study information with family members (optional).

It is expected that about 1500 people will take part in this research study. Participants will be in this study until it closes or the participant withdraws consent.

The National Cancer Institute is providing funding for part of this study and is considered a study sponsor. They will require that some of the genetic information be made available to the research community without personal identifying information.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a TP53 pathogenic or likely pathogenic variant identified in blood or saliva,
* Individuals with variants of uncertain significance in TP53 may be eligible at the PI's discretion,
* Blood relatives of individuals with a TP53 variant, who may be presumed obligate carriers or healthy controls,
* Individuals who meet Classic or Chompret LFS criteria whether or not they have a TP53 gene variant,
* Individuals may enroll their deceased relatives in the study.
* Individuals with a known TP53 variant that is not LFS, but rather ACE, CHIP, or mosaicism.
* Individuals participating in other LFS studies can still enroll in LiFT UP. Investigators may be collaborators.

Exclusion Criteria:

* Individuals who decline to sign consent
* Individuals who are unable to give consent or assent and are without a designated healthcare proxy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with a TP53 gene variant identified in blood or saliva
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Repository of specimens and data | 5 years or Study closure
  Examine accuracy of family history and the extent to which families meet various published Li-Fraumeni family criteria or assess for de-novo mutations using descriptive statistics. Exact binomial confidence limits for percents will be calculated at 95% coverage. Tests of difference between >2 groups for binary variables will use the Fisher exact test.

SECONDARY OUTCOMES:
Estimation of Cancer Risks in TP53 mutation carriers | 5 years or Study closure
  Estimate the frequency in ExAc as a population rate and calculate a standardized risk ratio as the ratio of the prevalence of mutations in a given cancer type compared to that in ExAc. P-values and 95% confidence intervals will be calculated assuming the observed number of mutations follows a Poisson distribution with mean equal to the expected value calculated from the ExAC observed frequency.
Modified segregation analysis | 5 years or Study closure
  For each dataset, the following analyses will be performed using MENDEL: a) the relative risk (RR) across age groups is assumed to be constant; b) the RR is assumed to be a continuous, piece wise linear function of age which was constant before age 40 years and after age 60 years, and linear between ages 40 and 60 years
Estimation of risk for the more commonly occurring cancers associated with inherited TP53 mutations | 5 years or Study closure
  P-values and 95% confidence intervals will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Judy E Garber, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Judy E. Garber, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] de Andrade KC, Lee EE, Tookmanian EM, Kesserwan CA, Manfredi JJ, Hatton JN, Loukissas JK, Zavadil J, Zhou L, Olivier M, Frone MN, Shahzada O, Longabaugh WJR, Kratz CP, Malkin D, Hainaut P, Savage SA. The TP53 Database: transition from the International Agency for Research on Cancer to the US National Cancer Institute. Cell Death Differ. 2022 May;29(5):1071-1073. doi: 10.1038/s41418-022-00976-3. Epub 2022 Mar 29. No abstract available. PMID 35352025